CLINICAL TRIAL: NCT02655211
Title: Laser Induced Bioengineered Remodeling of Thermally Injured Skin Trial: The Sequential Multiple Assignment Randomized Trial (SMART) Approach to Treatment of Hypertrophic Burn Scars
Brief Title: Laser Induced Bioengineered Remodeling of Thermally Injured Skin Trial
Acronym: LIBERTI
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to staff shortages we are closing the study.
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13-0735
Record Dates: First submitted 2014-11-12; First posted 2016-01-13 (Estimated); Last update posted 2017-04-17 (Actual); Status verified 2017-04

CONDITIONS: Hypertrophic Scars
MeSH Terms: conditions — Cicatrix, Hypertrophic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (12):
- CO2-CO2-Med (Active Comparator): Participants will receive two blocks of CO2 laser treatment, followed by one block of usual care.
  Interventions: Procedure: CO2 laser treatment; Other: Usual care
- Med-CO2-CO2 (Active Comparator): Participants will receive one block of usual care, followed by two blocks of CO2 laser therapy.
  Interventions: Procedure: CO2 laser treatment; Other: Usual care
- CO2-Med-CO2 (Active Comparator): Participants will receive one block of CO2 laser therapy, one block of usual care, and finally one more block of CO2 laser therapy.
  Interventions: Procedure: CO2 laser treatment; Other: Usual care
- PDL-PDL-MED (Active Comparator): Participants will receive two blocks of PDL laser therapy, followed by one block of usual care.
  Interventions: Procedure: PDL laser treatment; Other: Usual care
- Med-PDL-PDL (Active Comparator): Participants will receive one block of usual care, followed by two blocks of PDL laser therapy.
  Interventions: Procedure: PDL laser treatment; Other: Usual care
- PDL-Med-PDL (Active Comparator): Participants will receive one block of PDL laser therapy, followed by one block of usual care, followed by one block of PDL laser therapy.
  Interventions: Procedure: PDL laser treatment; Other: Usual care
- PDL-CO2-Med (Active Comparator): Participants will receive one block of PDL laser therapy, followed by one block of CO2 laser therapy, followed by one block of usual care.
  Interventions: Procedure: CO2 laser treatment; Procedure: PDL laser treatment; Other: Usual care
- CO2-PDL-Med (Active Comparator): Participants will receive one block of CO2 laser therapy, followed by one block of PDL laser therapy, followed by one block of usual care.
  Interventions: Procedure: CO2 laser treatment; Procedure: PDL laser treatment; Other: Usual care
- Med-PDL-CO2 (Active Comparator): Participants will receive one block of usual care, followed by one block of PDL laser therapy, followed by one block of CO2 laser therapy.
  Interventions: Procedure: CO2 laser treatment; Procedure: PDL laser treatment; Other: Usual care
- Med-CO2-PDL (Active Comparator): Participants will receive one block of usual care, followed by one block of CO2 laser therapy, followed by one block of PDL laser therapy.
  Interventions: Procedure: CO2 laser treatment; Procedure: PDL laser treatment; Other: Usual care
- PDL-Med-CO2 (Active Comparator): Participants will receive one block of PDL laser therapy, followed by one block of usual care, followed by one block of CO2 laser therapy.
  Interventions: Procedure: CO2 laser treatment; Procedure: PDL laser treatment; Other: Usual care
- CO2-Med-PDL (Active Comparator): Participants will receive one block of CO2 laser therapy, followed by one block of usual care, followed by one block of PDL laser therapy.
  Interventions: Procedure: CO2 laser treatment; Procedure: PDL laser treatment; Other: Usual care

INTERVENTIONS:
Procedure: CO2 laser treatment — Surgical treatment using fractionated ablative carbon dioxide laser (CO2)
  Arms: CO2-CO2-Med; CO2-Med-CO2; CO2-Med-PDL; CO2-PDL-Med; Med-CO2-CO2; Med-CO2-PDL; Med-PDL-CO2; PDL-CO2-Med; PDL-Med-CO2
Procedure: PDL laser treatment — Surgical treatment using flashlamp-excited pulsed dye laser (PDL)
  Arms: CO2-Med-PDL; CO2-PDL-Med; Med-CO2-PDL; Med-PDL-CO2; Med-PDL-PDL; PDL-CO2-Med; PDL-Med-CO2; PDL-Med-PDL; PDL-PDL-MED
Other: Usual care — Usual care (i.e., non-surgical) therapy (compression garments, massage, physical therapy, silicone gel sheeting)

SUMMARY:
This study will evaluate the efficacy of pulsed dye laser (PDL) and carbon dioxide (CO2) laser in conjunction with usual care (MED) for the treatment of hypertrophic burn scars and will determine the optimal sequence and timing of lasers and usual care.

DETAILED DESCRIPTION:
The investigator will compare usual care (MED), which will be offered to all patients, to two types of laser treatment (PDL and CO2), which the investigators hypothesize to be beneficial. The timing and sequence of therapy will be randomized, but all patients will receive some form of laser treatment. If the investigators simply stopped at the end of Aim 1, the investigators would complete a traditional randomized control trial (RCT), with some patients potentially receiving laser treatment. However, the investigators are interested in determining whether the sequence of laser treatments is beneficial; therefore, the investigators will be employing a sequential multiple assignment randomized trial (SMART) design. Because of the nature of the study and SMART design, the investigators will offer all patients some form of laser therapy.

ELIGIBILITY:
Inclusion Criteria:

* have a burn injury which will be at least 6 months old at the time of first treatment,
* have one or more symptomatic burn scars (with at least one or more symptoms such as erythema, pruritus, surface irregularity, or tightness not caused by a contracture that would be better served with surgical treatment),
* desire laser treatment,
* be at least 6 months of age at the time of treatment,
* agree to have no aesthetic treatments for their burn scars, such as peels or fillers, until they have completed the study (two-year period),
* agree to be randomized into one of the study's treatment conditions,
* agree to return for all treatment and follow-up visits for the two-year study period,
* agree to refrain from participating in any other treatment-oriented clinical trial for the duration of this study, and
* be able and willing to follow the protocol requirements.

Exclusion Criteria:

* be women who are pregnant or planning to become pregnant during the study,
* have had any previous laser treatment of their burn scars,
* have open wounds that are not re-epithelialized in the areas of proposed study treatment,
* be taking systemic steroids or immunosuppression medication,
* have a connective tissue disorder,
* be receiving or planning to receive chemotherapy or radiation during the study,
* be medically unable to tolerate anesthesia, or
* have other conditions that in the opinion of the investigators or clinicians may affect participant safety or compromise study objectives.

Ages: 6 Months to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-12; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Change in Hypotrophic scar score on the Vancouver Scar Scale (VSS) from baseline to three month visit | Baseline and 3 months

SECONDARY OUTCOMES:
Long-term hypotrophic scar score on VSS | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Scott Hultman, MD, Principal Investigator — UNC-Chapel Hill